CLINICAL TRIAL: NCT06965751
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of PDI204 as Intravenous Infusion or Intramuscular Injection in Healthy Participants
Brief Title: A Study on the Effects in Healthy People of a New Drug Called PDI204 for Treating COVID-19
Acronym: PHONIC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Nucleus Network Ltd (Other); Syneos Heath (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UoM-01-PDI204
Record Dates: First submitted 2025-04-29; First posted 2025-05-11 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; Phase 1; monoclonal antibody; healthy volunteers
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): PDI204 (anti SARS-CoV-2 spike proteinmonoclonal antibody) adminstered as a single intravenous or intramuscular dose
  Interventions: Drug: PDI204
- Placebo (Placebo Comparator): 0.9% saline administered as a single intravenous or intramuscular dose
  Interventions: Other: 0.9 % saline

INTERVENTIONS:
Drug: PDI204 — PDI204 is a fully human, immunoglobulin G1 (IgG1) monoclonal antibody (mAb) directed against the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein
  Arms: Active
Other: 0.9 % saline — 0.9% saline used as placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if a new drug called PDI204, developed for treating or preventing COVID-19, is safe and well-tolerated in healthy volunteers. This is a first-in-human study. The main questions it aims to answer are:

Is PDI204 safe and well-tolerated in healthy people? How long for and how does the body interact with PDI204?

Researchers will compare side effects in people who receive PDI204 and in those who receive a placebo (a look-alike substance that contains no drug) to see if and how many side-effects there are with PDI204. Researchers will also measure how long PDI204 can be detected in the blood.

Participants will be asked to receive a single dose of PDI204. Participants will have to stay in the clinical center for the day of receiving the dose of PDI204 and will be discharged the next day. Participants will then need to come back to the clinical center for study visits on days 3, 5, 7 (+/-1), 15 (+/-1), 30 (+/-3), 60 (+/-3) and 90 (+/-7).

DETAILED DESCRIPTION:
"A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (SAD) of PDI204 as Intravenous Infusion or Intramuscular Injection in Healthy participants" will be a single center, Phase 1, randomized, double-blind, placebo controlled, sequential single ascending dose (SAD) study evaluating the safety, tolerability, and pharmacokinetics (PK) of PDI204 via a single intravenous (IV) or intramuscular (IM) dose in healthy adult participants. The study will also assess the incidence and impact of antidrug antibodies (ADAs) on PK parameters and evaluate SARS-CoV-2 neutralizing antibody (NAb) levels over time. The study will consist of a single part with 4 cohorts: 3 sequential cohorts receiving IV administration (Cohorts 1-3) in an ascending dose manner, and one cohort receiving IM administration (Cohort 4), which may partially or fully overlap with the first 3 cohorts. Each cohort will include 8 participants (6 participants receiving the active drug and 2 participants receiving the placebo), for a total of 32 participants. The study will include a screening visit from Day -28 to Day -2. Eligible participants will be admitted to the clinical site on Day 1 and will be discharged on Day 2 following the completion of all required assessments. Participants will return to the clinical site for follow-up visits on Days 3, 5, 7 (+/-1), 15 (+/-1), 30 (+/-3), 60 (+/-3) and 90 (+/-7). The total duration of study participation for each participant from screening through the study exit is anticipated to be approximately 118 days. A staggered dosing schedule will be used for dosing of each cohort and will include 2 sentinel participants (1 active and 1 placebo) dosed initially, and the remaining 6 participants dosed at least 24 hours later in Cohorts 1a, 2a and 3a (IV administration); and at least 48 hours later in Cohort 2b (IM administration). The planned dose range for IV administration (Cohorts 1-3) is anticipated to be from 200 to 1200 mg, while a single 300 mg dose is planned for IM administration (Cohort 4).Following completion of each dose level, a Safety Review Committee (SRC) will review the safety and tolerability data, as well as available PK data, in order to make decisions whether to escalate to the next dose level, decrease the next dose level, repeat a dose level, or to not evaluate any additional dose. Additionally, the SRC may extend the duration of the IV infusion (Cohorts 1-3) if necessary to improve participant safety or tolerability.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, ≥18 and ≤65 years of age, with BMI >18.5 and <32.0 kg/m2. 2. Healthy as defined by:

  1. The absence of clinically significant illness and surgery within 4 weeks prior to study drug administration.
  2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease. Fully resolved basal cell carcinoma (BCC) and squamous cell carcinoma (SCC) are acceptable.

     3. Females of non-childbearing potential must be:

  <!-- -->

  1. post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented FSH levels 40 mIU/mL or greater; or
  2. surgically sterile (bilateral oophorectomy or hysterectomy) at least 3 months prior to dosing.

     4. Sexually active females of childbearing potential and non-sterile males must be willing to use an acceptable contraceptive method throughout the study as detailed in section 8.1.

     5. Male participants must be willing not to donate sperm for 90 days and female participants must be willing not to donate eggs for 30 days after dosing.

     6. Willing to abstain from alcohol, tobacco, and illicit drug use for 48 hours prior to admission to the CRU (Day -1) and during the inpatient period.

     7. Non-tattooed, clear injection site (i.e., absence of dermatologic conditions, such as scarring or rash, that may impact the ability to assess injection site reactions) suitable for IV or IM injection and monitoring in the opinion of the Investigator.

     8. Able to understand the study procedures and provide signed informed consent to participate in the study

     Exclusion Criteria:
     1. Any clinically significant abnormal finding at physical examination.
     2. Clinically significant abnormal laboratory test results or positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody, or QuantiFERON®-TB test at screening. Per Investigator's discretion, a single repeat for safety laboratory assessment to confirm initial result and trending is allowed per investigator's discretion.
     3. Positive pregnancy test or lactating female participant.
     4. Positive urine drug screen, or alcohol breath test.
     5. History of significant allergic reactions (e.g., anaphylactic reaction, hypersensitivity, angioedema) to any drug, in the opinion of investigator.
     6. Clinically significant ECG abnormalities or vital signs abnormalities (systolic BP lower than 90 or over 140 mmHg, diastolic BP lower than 40 or over 90 mmHg, HR less than 40 or over 100 bpm, or RR less than 10 or over 22 bpm) at screening.
     7. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening. per investigator's discretion, a single repeat for drug abuse urine test in the event of a false positive is allowed.
     8. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 14 units for women and 21 units for men of alcohol per week (1 unit = 200 mL of beer 5%, 83 mL of wine 12%, or 25 mL of distilled alcohol 40%).
     9. Participants who smoke more than 10 cigarettes per day or the equivalent per week.
     10. History of rare hereditary sucrose intolerance (e.g., genetic sucrose-isomaltase deficiency (GSID).
     11. History of a known or suspected respiratory system disorder including, but not limited to, cystic fibrosis, interstitial lung disease, reactive airway disease, emphysema, chronic bronchitis, pulmonary hypertension, COPD, or asthma (participants with childhood asthma can be included in the study).
     12. Diagnosis or suspected diagnosis of immunodeficiency or autoimmune diseases, or undergoing immunosuppressive therapy such as anticancer chemotherapy or radiotherapy before the study, or has received systemic corticosteroid treatment (topical corticosteroids are acceptable) within the past 120 days before dosing.
     13. Poor peripheral venous access for Cohorts 1a, 2a, and 3a.
     14. Fever (≥ 38.0°C) within 14 days before study drug administration.
     15. Positive Corona Virus Disease of 2019 (COVID-19) test at admission to the CRU.
     16. Vaccination (including COVID-19 vaccine) within 30 days prior to administration of PDI204.
     17. Known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to human proteins, mAbs or antibody fragments, or to any components of the formulation of PDI204 and its excipients used in this study.
     18. History of bleeding disorders or clotting disorders (e.g., hemophilia, thrombocytopenia) or those with a history of easy bruising or bleeding who may be at a higher risk for hematoma at the injection site.
     19. Participants who had close contact (without PPE) as defined by the Centers for Disease Control and Prevention (CDC) in the past 14 days to someone diagnosed with SARS-CoV-2 infection or COVID-19 within 10 days of the close contact. Participants may be rescreened after 14 days provided that they remain asymptomatic.
     20. Participants who have been infected by COVID-19, within 30 days prior to the drug administration.
     21. Has known active infection with influenza or other non-SARS-CoV-2 respiratory pathogen, confirmed by a diagnostic test.
     22. Previous infusion-related reaction, or severe adverse reaction following administration of a mAb.
     23. Use of medications within the timeframes specified in section 8.2.
     24. Participation in a clinical research study involving the administration of an investigational or marketed drug (including mAbs) or device within 30 days (or 5 half-lives since last receipt of an investigational drug, whichever is longer) prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
     25. Donation of serum within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 30 days prior to screening.
     26. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of a single IV or IM dose of PDI204 in healthy adult participants | Cumulative by Day 90
  Adverse events (AEs), serious adverse events (SAEs), vital signs measurements (blood pressure, heart rate, respiratory rate, and body temperature), 12-lead electrocardiogram (ECG) recordings, physical examinations, injection site reactions, and clinical laboratory test results, including hematology, biochemistry, and urinalysis; in the active arm compared with the placebo arm

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve to last observation (PDI204 pharmacokinetics: AUC0-t: time-averaged concentration ) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  AUC0-t: Area under the concentration-time curve from time zero until the last observed concentration
Area under the serum concentration versus time curve to infinity (PDI204 pharmacokinetics: time-averaged concentration to infinity, AUC0-inf) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  AUC0-inf: Area under the concentration-time curve from time zero to infinity (extrapolated)
Residual area (PDI204 pharmacokinetics; % of time-averaged concentration due to extrapolation) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  Residual area: Percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity, calculated as [1 - (AUC0-t/AUC0-inf)] x 100
Peak serum concentration (PDI204 pharmacokinetics: Cmax ) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  Cmax: Maximal observed concentration
Time of peak serum concentration (PDI204 pharmacokinetics: Tmax) | Day 1 - 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  Tmax: Time when the maximal concentration is observed
Elimination half-life (PDI204 pharmacokinetics:T 1/2 el ) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  T½ el: Terminal elimination half-life
Elimination rate constant (PDI204 pharmacokinetics: K el ) | Day 1 - predose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  K el: Terminal elimination rate constant
Clearance (PDI204 pharmacokinetics: Cl/F) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  Cl/F: Apparent clearance
Volume of distribution (PDI204 pharmacokinetics: Vz/F) | Day 1 - pre-dose, 30 minutes, 4 hours, 8 hours, 12 hours; Days 2, 3, 5, 7, 14, 30, 60 and 90
  In serum:
  Vz/F: Apparent volume of distribution
Incidence of anti-drug antibodies (ADAs) | Day 30
  Incidence of ADAs
Serum PK parameters with and without ADAs | Day 90
  Comparison of serum PK parameters for participants with versus without ADAs.
Changes in SARS-CoV-2 neutralising antibody (NAb) levels | Days 30 and 90
  Changes in SARS-CoV-2 NAb levels in serum and saliva from baseline
Incidence of anti-drug antibodies (ADAs) | Day 90
  Incidence of ADAs

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kent, PhD, MD, Principal Investigator — University of Melbourne
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie any published results, after deidentification (text, tables, figures, and appendices) will be shared. The Study Protocol and Informed Consent Form will also be made available. These data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee, for the purpose of participant data meta-analysis. The data will be available 3 months after publication and ending 5 years following publication. Proposals should be directed to Professor Stephen Kent (skent@unimelb.edu.au). To gain access to the data, requestors will need to sign a data sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available 3 months after publication and ending 5 years following publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee, for the purpose of participant data meta-analysis. Proposals should be directed to Professor Stephen Kent (skent@unimelb.edu.au). To gain access to the data, requestors will need to sign a data sharing agreement.